CLINICAL TRIAL: NCT01775293
Title: A Multi Center, Non-comparative Clinical Study to Evaluate the Correction of Facial Wrinkles and Folds and Safety After Rhytidectomy Using Non-absorbable Mesh(RPM)
Brief Title: Clinical Trial to Evaluate the Efficacy and Safety in Nasolabial Fold After Rhytidectomy Using Non-absorbable Mesh
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: D.med (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E-1209-170-002; 06-2012-208 (Other: Seoul National University Bundang Hospital)
Record Dates: First submitted 2013-01-22; First posted 2013-01-24 (Estimated); Last update posted 2014-01-07 (Estimated); Status verified 2014-01

CONDITIONS: Nasolabial Fold
Keywords: Non-absorbable polypropylene mesh; WSRS; Rhytidectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Non-absorbable polypropylene mesh (Experimental): 2 step procedures
  * first step is insertion of Non-absorbable polypropylene mesh under the facial skin
  * second step is pulling of Non-absorbable polypropylene mesh after 3 weeks of 1 step
  Interventions: Device: Non-absorbable polypropylene mesh

INTERVENTIONS:
Device: Non-absorbable polypropylene mesh — 2 step procedures
  * first step is insertion of Non-absorbable polypropylene mesh under the facial skin
  * second step is pulling of Non-absorbable polypropylene mesh after 3 weeks of 1 step

SUMMARY:
The aim of this study is to evaluate the efficacy and safety of the investigational device, RPM,non-absorbable polypropylene mesh made by D Med, in correction of Nasolabial fold.

Study hypothesis

* level of significance: alpha=0.05( two-side)
* power of test: (power= 1-beta),power=0.08
* H0: P equals P0
* H1: P unequals P0
* The difference between the changes in the WSRS(Wrinkle Severity Rating Scale) of the pre and post rhytidectomy from baseline at 7week after administration is 0.237( P-P0= 0.237)

DETAILED DESCRIPTION:
1. Benefits

* enhancing self-satisfaction and quality of life by improving skin elasticity and correcting folds in the nasolabial fold area 2. Risks
* erythema, swelling, pain and redness in the facial area generally resolve in 1 week 3.Duration of study
* entire duration: approximate 36weeks
* Follow-up period: 7 weeks
* Enrollment period: 12 weeks 4. study design
* 2 step operation process

  * First step- insert polypropylene mesh under the skin
  * Second step- pull the polypropylene mesh 3 weeks later

ELIGIBILITY:
Inclusion Criteria:

* Subjects who had soft tissue sagging around nasolabial fold
* Female aged between 30 and 65, having grade 3 or 4 of nasolabial fold as Wrinkle severity Rating Scale(WSRS)
* Subjects who voluntary decided to participate in the study and signed the informed consent

Exclusion Criteria:

* Subjects who have a skin disease on the face
* Subjects who have severe facial skin disease
* Subjects who are constantly taking anti-coagulants including aspirin
* Subjects who have too thin or thick skin
* Subjects who have a systemic disease such as uncontrolled high blood pressure, diabetes, heart disease
* Subjects who had an allergy to non-absorbable material.
* Subjects who are taking immune suppressants
* General weakness status
* Pregnant or lactating women
* Subjects who have an asthma, cancer, AIDS, Cystic fibrosis, Immobility cilia syndrome, leukopenia, Immunoglobulin deficiency, active infectious disease, serious liver or renal disease,
* Subjects who had a history of dermal augmentation surgery with permanent implants(e.g. silicone, Softform®)on the face
* Subjects who participated in other clinical trial within 30 days from screening

Ages: 30 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2013-01; Primary Completion 2013-12 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
The change in the WSRS(Wrinkle Severity Rating Scale) of the pre and post rhytidectomy from baseline at 7week after administration | change in the WSRS from baseline at7 week
  The efficacy is assessed by the severity of the fold determined by the WSRS assessed by the investigator with photos WSRS(Wrinkle Severity Rating Scale)is be evaluated from 1 to 5 according to the severity of wrinkles
  (1= no visible fold, 5= extremely deep and long fold)

SECONDARY OUTCOMES:
The changes in the satisfaction of the pre and post rhytidectomy from baseline at 7week after administration | Changes Satisfaction from baseline at 7week
  The changes in the satisfaction(VAS-visual analog scale) of the pre and post rhytidectomy from baseline at 7week after administration VAS(visual analog scale)is to be evaluated from 0 to 100 by the participant ( 0= no wrinkle, 100= severe wrinkle)

CONTACTS AND LOCATIONS:
Overall Officials: Chanyeong Heo, Master, Principal Investigator — Seoul National University Hospital
Locations (1):
- Korea University Anam Hospital, Seoul, Seongbukgu/Seoul, South Korea